CLINICAL TRIAL: NCT05186051
Title: A Phase 2a, Prospective, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZYIL1 in Subjects With Cryopyrin Associated Periodic Syndromes (CAPS)
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZYIL1 in Subjects With Cryopyrin Associated Periodic Syndromes (CAPS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYIL1.21.001
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2021-12

CONDITIONS: Cryopyrin Associated Periodic Syndrome
Keywords: NLRP3; NLPR3 Inflammasone inhibitor
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes | interventions — ZYIL1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZYIL1 Capsule (Experimental): subject will receive 50 mg twice daily (BD) dose for 7 days
  Interventions: Drug: ZYIL1 capsule

INTERVENTIONS:
Drug: ZYIL1 capsule — NLRP3 inflammasome inhibitor

SUMMARY:
ZYIL1 is expected to show benefit in patients with CAPS. The present study aims to determine the safety, tolerability, pharmacokinetics, and pharmacodynamics of ZYIL1 when administered to subjects with CAPS.

DETAILED DESCRIPTION:
This is a phase 2a, prospective, open-label study. Primary objective of the study is to determine safety and tolerability profile of twice daily oral administration of ZYIL1 administered for 7 days. The study will be conducted in 3 subjects having CAPS as per eligibility criteria. The study will be divided in three periods: Screening Period; Run-in Period and Study Period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a confirmed diagnosis of CAPS (FCAS, NOMID, or MWS) aged 18 to 75 years inclusive at screening A confirmed diagnosis of CAPS comprises the following:

   1. Subject has previously experienced at least 2 typical clinical symptoms of CAPS (may include urticarial skin rash, myalgia, arthralgia, recurrent fever, fatigue/malaise, headache, conjunctivitis, and any other autoinflammatory symptom); and
   2. Documented verification of a genetic mutation in NLRP3.
2. Positive response of ZYIL1 in inhibiting secreted IL-1β from peripheral blood mononuclear cells isolated from the subject's blood treated with LPS ex vivo showing half maximal inhibitory concentration below 500 nM.
3. Subject must be willing to discontinue current anti-IL-1 treatment prior to study drug dosing if applicable.
4. Subject must demonstrate flaring of CAPS de novo or after discontinuation of anti-IL-1 inhibitor treatment. Flaring is defined as worsening of disease activity as per physician global assessment of disease activity with elevation of CRP (>2 x upper limit of normal [ULN]).
5. Subject must have a body mass index (BMI) between ≥18.0 and ≤38.0 kg/m2 at Screening.
6. Female subject of reproductive age must be non-pregnant and non-lactating, and must use an acceptable, highly effective contraception from screening until 1 month after the last dose of study drug.
7. Male subject must be willing to use contraception and must not donate sperm for at least 90 days after the last dose of study drug.

Exclusion Criteria:

1. Any severe, progressive, or uncontrolled medical condition within the past 3 months that might have impact on the clinical trial as per the investigator's discretion.
2. Use of any investigational drug or investigational medical device or participation in other clinical study within 4 weeks prior to Screening or 5 half- lives of the product (whichever is longer).
3. Any clinically significant laboratory or ECG findings during the screening in the opinion of the Investigator.
4. Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m2, as measured by the Cockcroft-Gault equation at screening
5. Total bilirubin above upper limit of normal (ULN) or AST(SGOT)/ALT(SGPT) > 1.5 times of ULN at screening
6. QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 msec at screening
7. History of clinically significant hypersensitivity, intolerance, or allergies, as determined by the investigator.
8. History of fever, cough or any other active systemic infections within 2 weeks prior to receiving study drug.
9. History or presence of alcohol abuse (alcohol consumption more than 40 g/4 units/4standard drinks per day), or drug habituation, or any prior intravenous usage of an illicit substance
10. Surgery within last 3 months or planned major surgery within next 3 months from the date of screening (other than minor cosmetic surgery and minor dental surgery).
11. Subjects who have donated one unit (490 mL) of blood in the past 3 months.
12. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes including St John's Wort within 4 weeks prior to receiving study drug and up to end of study. Use of such medication will be considered on a case-by-case basis as per the opinion of the investigator and/or independent medical monitor, or use of grapefruit or similar substances (Seville oranges or marmalade, grapefruit juice, grapefruit hybrids, pomelos, exotic citrus fruits or fruit juices) within 7 days prior to the Run-in period.
13. Use or intend to use any over-the-counter (vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) or prescription medications within 7 days or 5 half-lives (whichever is longer) prior to receiving study drug, with the exception of hormone replacement therapy and therapies for chronic stable diseases that have been stable for at least 30 days prior to screening and until Day 1, unless deemed acceptable by the investigator
14. History of or positive screening test for hepatitis C infection (defined as positive for hepatitis C virus antibody), hepatitis B infection (defined as positive for hepatitis B surface antigen), or human immunodeficiency virus I or II.
15. Female subjects who are pregnant, currently breastfeeding, or attempting to conceive.
16. Any disorder that, in the Investigator's opinion, may interfere with study compliance, such as significant mental, nervous disorder or other illness. In making this assessment, the Investigator must refer to the study information provided including the Investigator's Brochure.
17. Inability to be venipuncture or tolerate venous puncture.
18. Any condition or abnormal baseline findings that in investigator's judgment might increase the risk to the subject or decrease the chance of obtaining satisfactory data needed to obtain the objective of the study.
19. Other unspecified reasons that, in the opinion of the investigator make the subject unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse event of ZYIL1 | Baseline to Day 7
  The Common Terminology Criteria for Adverse Event (CTCAE) (Version 5.0 or higher) system will be used for reporting and grading

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Pre-dose to Day 7
  Blood samples will be withdrawn on Day 1 and Day 7 to evaluate maximum concentration
To evaluate disease activity scores based on 5 point physician and patient global assessment over 7 days treatment of ZYIL1 | Baseline to Day 10
  Physician global assessment on 5 point scale score will be taken
Time to reach maximum concentration (Tmax) | Pre-dose to Day 7
  Blood samples will be withdrawn on Day 1 and Day 7 to evaluate Time to reach maximum concentration
Area under the curve for dosing interval(12 hours) AUCtau | Pre-dose to Day 7
  Blood samples will be withdrawn on Day 1 and Day 7 to evaluate AUCtau
Change in WBC count | Baseline to Day 10
  Blood samples will be collected from pre-dose till Day 10 to evaluate the change
Change in IL-1β | Baseline to Day 10
  Blood samples will be collected from pre-dose till Day 10 to evaluate the change
Change in Serum amyloid protein A | Baseline to Day 10
  Blood samples will be collected from pre-dose till Day 10 to evaluate the change
Change in IL-6 | Baseline to Day 10
  Blood samples will be collected from pre-dose till Day 10 to evaluate the change
Change in CRP | Baseline to Day 10
  Blood samples will be collected from pre-dose till Day 10 to evaluate the change

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deven Parmar, MD, Study Director — Cadila Healthcare Ltd.
Locations (1):
- Department of Clinical Immunology and Allergy, Adelaide, Australia